CLINICAL TRIAL: NCT01837810
Title: NSAID Post-Tonsillectomy Hemorrhage: A Randomized, Double-Blinded Controlled Noninferiority Trial
Brief Title: Safety Study of Post Tonsillectomy Ibuprofen Use in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); Blanchfield Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gregory R. Dion, MD, MS, CPT, MC, USA, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 384409
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Secondary Post Tonsillectomy Hemorrhage; Primary Post Tonsillectomy Hemorrhage
Keywords: Post tonsillectomy hemorrhage; post operative hemorrhage; complications; tonsillectomy
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Experimental): 800mg ibuprofen every 8 hours prn pain.
  Interventions: Drug: Ibuprofen
- Methylcellulose Powder (Placebo Comparator): Subjects receive inert methylcellulose powder as placebo

INTERVENTIONS:
Drug: Ibuprofen — 800mg every 8 hours as needed for pain
  Other Names: Advil; Motrin
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to determine if ibuprofen use after electrocautery tonsillectomy increases the post-tonsillectomy hemorrhage rate.

Hypothesis: Use of ibuprofen does not increase the post-tonsillectomy hemorrhage rate.

Primary outcome: Rate of tonsillar hemorrhage following adult tonsillectomy in those receiving narcotic pain medications plus ibuprofen compared to those receiving narcotics alone.

Secondary outcome: Determine whether ibuprofen, a non-steroidal anti-inflammatory drug (NSAID), decreases post tonsillectomy pain, narcotic pain medication use, or cost of pain management.

DETAILED DESCRIPTION:
Tonsillectomy is common procedure associated with significant post-operative pain typically managed by narcotic pain medication. Narcotics, however, can have inherent unwanted side effects such as respiratory depression. In fact, a recent U.S. Food and Drug Administration (FDA) warning has reported deaths from respiratory distress that were associated with use of codeine in children after tonsillectomy. Finding alternative pain management regimens therefore is essential in post-tonsillectomy care. Non-steroidal anti-inflammatory (NSAID) medications may provide an effective alternative to narcotics, but use of NSAIDs routinely after tonsillectomy has been limited due to concern for theoretical increased risk of post-operative bleeding, This is likely true for NSAIDs such as aspirin. NSAIDs such as ibuprofen, however, are believed to have no greater risk of bleeding than baseline, but this has not been proven. Recent, well-designed, prospective pediatric studies have demonstrated effective analgesia improvement with the addition of non-steroidal anti-inflammatory drugs such as ibuprofen to post-operative pain management regimens, and no increased rate of post-surgery bleeding. This has not adequately been studied in adults but could provide many patients significant pain relief in the post-operative period if it is shown to not increase post tonsillectomy hemorrhage rates, as already demonstrated in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or older
* Scheduled for tonsillectomy

Exclusion Criteria:

* Prisoners
* Pregnancy
* Allergy to ibuprofen
* History of vasculopathy to include Lupus or Wegener's or Disseminated Intravascular Coagulation (DIC)
* Any other bleeding disorder to include Von Willebrand Disease and others
* Active Neoplasm of any kind
* Tonsillectomy in combination with any sleep surgical procedure or palatal procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
clinically defined tonsil bleed rate (percentage) | 2 weeks
  A post tonsillectomy hemorrhage/bleed, for the purposes of this study, is defined as a postoperative bleed requiring anything more than medicinal intervention (cauterization of any kind, suture, evaluation in operating room).

SECONDARY OUTCOMES:
Hospital readmission rate (percentage) | 2 weeks
Subclinical (not requiring intervention) subjectively reported tonsil bleed rate (percentage) | 2 weeks
  Subjects will report on followup survey if they had post operative oral bleeding more than streaked blood in their spit for which they did not go to the hospital or clinic for treatment of.
Pain scale rating | 2 Weeks
  Subjects will answer a visual analog scale (VAS) Pain scale for days 1, 3, 7, and 14 after tonsillectomy.
Nausea Scale | 2 weeks
  Subjects will answer a VAS nausea scale for days 1, 3, and 7 after tonsillectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory R Dion, MD, MS, Principal Investigator — San Antonio Military Medical Center
Locations (3):
- United States (3):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas
  - Madigan Army Medical Center, Tacoma, Washington